CLINICAL TRIAL: NCT03712631
Title: Ridge Augmentation in Atrophic Posterior Mandible Using Tunneling Technique With Anorganic Bovine Bone-Derived Mineral Mixed With Particulated Autogenous Bone Chips With and Without Collagen Membrane
Brief Title: Ridge Augmentation in Posterior Mandible Using Tunneling Technique With Amix of Autogenous Bone and Xenograft With and Without Collagen Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, haytham mohamed ahmed ibrahim, dr, Cairo University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: augmentation tunneling tech
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Alveolar Ridge Augmentation
Keywords: tunneling technique; collagen membrane; tunnel; augmentation; horizontal ridge augmentation; bone graft; ridge augmentation; posterior mandible

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bone without a collagen membrane (Active Comparator): not covering bone with collagen membrane
  Interventions: Procedure: tunneling technique bone augmentation
- bone with collagen membrane (Experimental): covering bone with collagen membrane
  Interventions: Procedure: tunneling technique bone augmentation

INTERVENTIONS:
Procedure: tunneling technique bone augmentation — horizontal ridge augmentation using mixture of xenograft,autogenous bone

SUMMARY:
aim Evaluation of the amount of bone gain following Ridge augmentation using tunneling technique in atrophic posterior mandibular ridges using anorganic bovine bone derived mineral mixed with particulated autogenous bone chips with collagen membrane

DETAILED DESCRIPTION:
Bone grafting before implant placement has become a routine procedure over the last 20 years. A 5-year survival rate of up to98.3% for implants placed in grafted bone has been reported.

Autologous bone grafts are considered the gold standard.However, the success rate of the grafting procedure may beinfluenced by various risk factors.

A particular challenge isposed by an extensive graft of the alveolar ridge, with relativelyhigh complication rates of up to 20% being reported, mostcommonly dehiscence. More serious complications such asdehiscence or mobilization of the graft were observed in one third of smokers compared to a complication rate of only 7.7%for non-smokers. Complications such as flap necroses, dehiscenceand resorption are frequently soft-tissue complications.

A tension-free wound closure is a key factor in the successof bone grafts. Periosteal incisions are a common techniquefor flap extension. However, too many relief incisions in the periosteum may also result in an excessively thin or stretched wound flap.

This type of soft-tissue management may result in perforation or flap necrosis above the bone graft.

In 1987 Härle reported on a tunneling access in connectionwith a technique for preprosthetic jaw ridge grafting in the mandibular side-tooth region with bone replacement materials.

In the clinical experience of the authors the use of a tunneling technique for preparation without a crestal incision can present an alternative with autologous bone grafts to conventional surgical procedures with a trapezoid flap design.

ELIGIBILITY:
Inclusion Criteria:

* medically free,age 22:50 years, atrophic posterior mandibleClinical diagnosis of Alzheimer's Disease Must be able to swallow tablets

Exclusion Criteria:

smoking Insulin dependent diabetes Clinical diagnosis of Alzheimer's Disease Must be able to swallow tablets

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Height and width of bone gained | 4 months

SECONDARY OUTCOMES:
Bone area percentage | 4 months

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within 2 years

REFERENCES:
- [Background] Hasson O. Augmentation of deficient lateral alveolar ridge using the subperiosteal tunneling dissection approach. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Mar;103(3):e14-9. doi: 10.1016/j.tripleo.2006.10.019. Epub 2007 Jan 22. PMID 17241798
- [Background] Maestre-Ferrin L, Boronat-Lopez A, Penarrocha-Diago M, Penarrocha-Diago M. Augmentation procedures for deficient edentulous ridges, using onlay autologous grafts: an update. Med Oral Patol Oral Cir Bucal. 2009 Aug 1;14(8):e402-7. PMID 19415058
- [Background] de Macedo LG, de Macedo NL, do Socorro Ferreira Monteiro A. Fresh-frozen human bone graft for repair of defect after adenomatoid odontogenic tumour removal. Cell Tissue Bank. 2009 Aug;10(3):221-6. doi: 10.1007/s10561-008-9120-1. Epub 2009 Jan 9. PMID 19132551
- [Background] Khan SN, Cammisa FP Jr, Sandhu HS, Diwan AD, Girardi FP, Lane JM. The biology of bone grafting. J Am Acad Orthop Surg. 2005 Jan-Feb;13(1):77-86. PMID 15712985
- [Background] 9. Fonseca RJ, Powers MP, Dexter H. Oral and max¬illofacial surgery: Reconstructive and implant surgery. Philadelphia: WB Saunders Co. 2007; 7.
- [Background] Kent JN. Reconstruction of the alveolar ridge with hydroxyapatite. Dent Clin North Am. 1986 Apr;30(2):231-57. PMID 3009242
- [Background] Smiler D, Soltan M, Lee JW. A histomorphogenic analysis of bone grafts augmented with adult stem cells. Implant Dent. 2007 Mar;16(1):42-53. doi: 10.1097/ID.0b013e3180335934. PMID 17356371
- [Background] Rothstein SS, Paris DA, Zacek MP. Use of hydroxylapatite for the augmentation of deficient alveolar ridges. J Oral Maxillofac Surg. 1984 Apr;42(4):224-30. doi: 10.1016/0278-2391(84)90453-1. PMID 6323657
- [Background] Mehlisch DR, Taylor TD, Leibold DG, Hiatt R, Waite DE, Waite PD, Laskin DM, Smith ST. Collagen/hydroxylapatite implant for augmenting deficient alveolar ridges: twelve-month clinical data. J Oral Maxillofac Surg. 1988 Oct;46(10):839-43. doi: 10.1016/0278-2391(88)90046-8. PMID 2845038
- [Background] Williams CW, Meyers JF, Robinson RR. Hydroxyapatite augmentation of the anterior portion of the maxilla with a modified transpositional flap technique. Oral Surg Oral Med Oral Pathol. 1991 Oct;72(4):395-9. doi: 10.1016/0030-4220(91)90546-o. PMID 1656356
- [Background] Marshall SG. The combined use of endosseous dental implants and collagen/hydroxylapatite augmentation procedures for reconstruction/augmentation of the edentulous and atrophic mandible: a preliminary report. Oral Surg Oral Med Oral Pathol. 1989 Oct;68(4 Pt 2):517-25; discussion 525-6. doi: 10.1016/0030-4220(89)90231-4. PMID 2559388
- [Background] Kfir E, Kfir V, Eliav E, Kaluski E. Minimally invasive guided bone regeneration. J Oral Implantol. 2007;33(4):205-10. doi: 10.1563/1548-1336(2007)33[205:MIGBR]2.0.CO;2. PMID 17912961
- [Background] Li J, Xuan F, Choi BH, Jeong SM. Minimally invasive ridge augmentation using xenogenous bone blocks in an atrophied posterior mandible: a clinical and histological study. Implant Dent. 2013 Apr;22(2):112-6. doi: 10.1097/ID.0b013e3182805bec. PMID 23344366
- [Background] Vanassche BJ, Stoelinga PJ, de Koomen HA, Blijdorp PA, Schoenaers JH. Reconstruction of the severely resorbed mandible with interposed bone grafts and hydroxylapatite. A 2-3 year follow-up. Int J Oral Maxillofac Surg. 1988 Jun;17(3):157-60. doi: 10.1016/s0901-5027(88)80021-3. PMID 2840471
- [Background] Block MS. Horizontal ridge augmentation using particulate bone. Atlas Oral Maxillofac Surg Clin North Am. 2006 Mar;14(1):27-38. doi: 10.1016/j.cxom.2005.11.004. No abstract available. PMID 16522508
- [Background] Block MS, Degen M. Horizontal ridge augmentation using human mineralized particulate bone: preliminary results. J Oral Maxillofac Surg. 2004 Sep;62(9 Suppl 2):67-72. doi: 10.1016/j.joms.2004.05.209. PMID 15332183
- [Background] Kuemmerle JM, Oberle A, Oechslin C, Bohner M, Frei C, Boecken I, von Rechenberg B. Assessment of the suitability of a new brushite calcium phosphate cement for cranioplasty - an experimental study in sheep. J Craniomaxillofac Surg. 2005 Feb;33(1):37-44. doi: 10.1016/j.jcms.2004.09.002. Epub 2005 Jan 11. PMID 15694148
- [Background] Flautre B, Maynou C, Lemaitre J, Van Landuyt P, Hardouin P. Bone colonization of beta-TCP granules incorporated in brushite cements. J Biomed Mater Res. 2002;63(4):413-7. doi: 10.1002/jbm.10262. PMID 12115749
- [Background] Penel G, Leroy N, Van Landuyt P, Flautre B, Hardouin P, Lemaitre J, Leroy G. Raman microspectrometry studies of brushite cement: in vivo evolution in a sheep model. Bone. 1999 Aug;25(2 Suppl):81S-84S. doi: 10.1016/s8756-3282(99)00139-8. PMID 10458282
- [Background] Heller AL, Heller RL, Cook G, D'Orazio R, Rutkowski J. Soft tissue management techniques for implant dentistry: a clinical guide. J Oral Implantol. 2000;26(2):91-103. doi: 10.1563/1548-1336(2000)0262.3.CO;2. PMID 11831336
- [Background] Heller AL, Heller RL. Tissue management protocol: "tunnel bone graft" technique. Dent Today. 2010 Nov;29(11):120, 122, 124. No abstract available. PMID 21133027
- [Background] Dahlin C, Gottlow J, Linde A, Nyman S. Healing of maxillary and mandibular bone defects using a membrane technique. An experimental study in monkeys. Scand J Plast Reconstr Surg Hand Surg. 1990;24(1):13-9. doi: 10.3109/02844319009004514. PMID 2389116
- [Background] Buser D, Dula K, Belser U, Hirt HP, Berthold H. Localized ridge augmentation using guided bone regeneration. 1. Surgical procedure in the maxilla. Int J Periodontics Restorative Dent. 1993;13(1):29-45. PMID 8330945
- [Background] Simion M, Baldoni M, Rossi P, Zaffe D. A comparative study of the effectiveness of e-PTFE membranes with and without early exposure during the healing period. Int J Periodontics Restorative Dent. 1994 Apr;14(2):166-80. PMID 7928132
- [Background] Machtei EE. The effect of membrane exposure on the outcome of regenerative procedures in humans: a meta-analysis. J Periodontol. 2001 Apr;72(4):512-6. doi: 10.1902/jop.2001.72.4.512. PMID 11338304
- [Background] Block MS, Kelley B. Horizontal posterior ridge augmentation: the use of a collagen membrane over a bovine particulate graft: technique note. J Oral Maxillofac Surg. 2013 Sep;71(9):1513-9. doi: 10.1016/j.joms.2013.05.015. PMID 23948364
- [Background] Deeb GR, Wilson GH, Carrico CK, Zafar U, Laskin DM, Deeb JG. Is the Tunnel Technique More Effective Than Open Augmentation With a Titanium-Reinforced Polytetrafluoroethylene Membrane for Horizontal Ridge Augmentation? J Oral Maxillofac Surg. 2016 Sep;74(9):1752-6. doi: 10.1016/j.joms.2016.04.031. Epub 2016 May 7. PMID 27240025
- [Background] Misch CM. Comparison of intraoral donor sites for onlay grafting prior to implant placement. Int J Oral Maxillofac Implants. 1997 Nov-Dec;12(6):767-76. PMID 9425757
- [Background] von Arx T, Hardt N, Wallkamm B. The TIME technique: a new method for localized alveolar ridge augmentation prior to placement of dental implants. Int J Oral Maxillofac Implants. 1996 May-Jun;11(3):387-94. PMID 8752560
- [Background] Chiapasco M, Abati S, Romeo E, Vogel G. Clinical outcome of autogenous bone blocks or guided bone regeneration with e-PTFE membranes for the reconstruction of narrow edentulous ridges. Clin Oral Implants Res. 1999 Aug;10(4):278-88. doi: 10.1034/j.1600-0501.1999.100404.x. PMID 10551070
- [Background] Harris RJ. Soft tissue ridge augmentation with an acellular dermal matrix. Int J Periodontics Restorative Dent. 2003 Feb;23(1):87-92. PMID 12617372
- [Background] Yan JJ, Tsai AY, Wong MY, Hou LT. Comparison of acellular dermal graft and palatal autograft in the reconstruction of keratinized gingiva around dental implants: a case report. Int J Periodontics Restorative Dent. 2006 Jun;26(3):287-92. PMID 16836171
- [Background] AlGhamdi AS, Buhite RJ. A new tunnel technique with acellular dermal matrix for soft tissue preparation prior to symphyseal block graft--a description of technique and case report. J Oral Implantol. 2008;34(5):274-81. doi: 10.1563/1548-1336(2008)34[275:ANTTWA]2.0.CO;2. PMID 19170294
- [Background] Lee CT, Hamalian T, Schulze-Spate U. Minimally invasive treatment of soft tissue deficiency around an implant-supported restoration in the esthetic zone: modified VISTA technique case report. J Oral Implantol. 2015 Feb;41(1):71-6. doi: 10.1563/AAID-JOI-D-13-00043. Epub 2013 Mar 19. PMID 23510339
- [Background] Cortellini P, Tonetti MS. A minimally invasive surgical technique with an enamel matrix derivative in the regenerative treatment of intra-bony defects: a novel approach to limit morbidity. J Clin Periodontol. 2007 Jan;34(1):87-93. doi: 10.1111/j.1600-051X.2006.01020.x. PMID 17243998
- [Background] Rothamel D, Schwarz F, Herten M, Ferrari D, Mischkowski RA, Sager M, Becker J. Vertical ridge augmentation using xenogenous bone blocks: a histomorphometric study in dogs. Int J Oral Maxillofac Implants. 2009 Mar-Apr;24(2):243-50. PMID 19492639
- [Background] Sammartino G, Pantaleo G, Nuzzolo P, Amato M, Riccitiello F. Minimally Invasive Approaches to Optimize Block Grafting: A Case Report. J Oral Implantol. 2016 Apr;42(2):176-9. doi: 10.1563/aaid-joi-D-14-00076. Epub 2014 Sep 18. No abstract available. PMID 25233065
- [Background] Misch CE, Dietsh F. Bone-grafting materials in implant dentistry. Implant Dent. 1993 Fall;2(3):158-67. doi: 10.1097/00008505-199309000-00003. PMID 8142935
- [Result] McAllister BS, Haghighat K. Bone augmentation techniques. J Periodontol. 2007 Mar;78(3):377-96. doi: 10.1902/jop.2007.060048. PMID 17335361